CLINICAL TRIAL: NCT07116798
Title: Investigation of the Effects of Different Upper Extremity Strengthening Exercises in Children With Unilateral Spastic Type Cerebral Palsy
Brief Title: Upper Extremity Strengthening Interventions in Children With UCP
Acronym: PNF vs PLY-UCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Gülsena Utku Umut, Assisstant Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: FTR-UCP-001
Record Dates: First submitted 2025-08-07; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Palsy (CP)
Keywords: cerebral palsy; upper extremity; strengthening
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF Group (Strengthening Based on Proprioceptive Neuromuscular Facilitation Patterns) (Experimental): The shoulder and scapular patterns listed below will first be taught to the child using the rhythmic initiation technique. Following instruction, the child will be asked to perform the patterns actively without resistance.
  Shoulder flexion - adduction - external rotation and shoulder extension - abduction - internal rotation (with the elbow extended) Shoulder extension - adduction - internal rotation and shoulder flexion - abduction - external rotation (with the elbow extended) In addition to the shoulder patterns, scapular patterns including anterior depression - posterior elevation and anterior elevation - posterior depression will also be performed with the same progression.
  Interventions: Other: Exercise
- Plyometric Group (Plyometric Exercises) (Experimental): Participants in the plyometric group will perform upper extremity plyometric exercises aimed at improving muscular power, neuromuscular control, and functional performance. The exercises will be selected to provide dynamic resistance and emphasize rapid stretch-shortening cycle movements of the upper limb. Training will be conducted using elastic bands, medicine balls, and body weight as appropriate to the child's developmental level and physical capacity. The exercise program will include progressive variations in terms of intensity, volume (sets and repetitions), and complexity over the intervention period, as detailed in the progression table. Rest intervals of no more than one minute will be allowed between sets. All exercises will be performed bilaterally and under the supervision of a physiotherapist to ensure proper technique and safety.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Strengthening Exercises Based on Proprioceptive Neuromuscular Facilitation Patterns
  Arms: PNF Group (Strengthening Based on Proprioceptive Neuromuscular Facilitation Patterns)
Other: Exercise — Plyometric Exercises
  Arms: Plyometric Group (Plyometric Exercises)

SUMMARY:
This study aims to compare the effects of two different upper extremity strengthening exercise approaches-bilateral strengthening exercises based on Proprioceptive Neuromuscular Facilitation (PNF) patterns and plyometric exercises-on muscle thickness, joint range of motion, muscle strength, and functional performance in children with unilateral spastic cerebral palsy (USCP). Although strengthening exercises targeting the affected upper limb in children with USCP have been investigated in numerous studies, to our knowledge, no previous research has directly compared the effects of bilateral PNF-based strengthening exercises and plyometric training. Incorporating PNF patterns into upper extremity rehabilitation programs has been previously recommended, and examining the efficacy of these exercises in comparison with plyometric training may contribute valuable insights to the literature and inform clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 5 and 12 years
* Diagnosed with unilateral spastic type cerebral palsy
* Classified as Level I or II according to the Gross Motor Function Classification System (GMFCS)
* Classified as Level I or II according to the Manual Ability Classification System (MACS)
* Upper extremity muscle tone ≤2 on the Modified Ashworth Scale
* Willing to suspend other upper extremity therapeutic interventions during the study period
* Able to cooperate and follow instructions provided by the researcher
* Voluntarily willing to participate in the study

Exclusion Criteria:

* History of any upper extremity surgery or Botulinum toxin (Btx) injection within the past 6 months
* Presence of an additional neurological disorder other than cerebral palsy
* Having visual and/or hearing impairments
* Having severe contractures that limit participation in functional activities

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-07-07 (Estimated)

PRIMARY OUTCOMES:
Muscle Thickness Measurement by Ultrasonography | Baseline and after 8-weeks
  Ultrasonographic measurements will be performed using the Esaote Mylab 60 device with a linear probe. Muscle thickness will be assessed in the upper trapezius, rhomboid major, anterior deltoid, lateral triceps brachii, long head of biceps brachii, extensor carpi radialis brevis, extensor digitorum communis, and flexor digitorum superficialis. Measurements will be taken with the elbow flexed at 70°, in standardized resting positions, with forearm in pronation or supination depending on the muscle group. To ensure reliability, three separate images per muscle will be taken, with the probe repositioned each time. Anatomical landmarks will be palpated and marked. Muscle thickness will be measured as the distance between the subcutaneous fat-muscle and muscle-bone interfaces.
Range of Motion Assessment | Baseline and after 8-weeks
  Joint range of motion (ROM) will be assessed before and after treatment using a universal goniometer. Active ROM measurements will include shoulder flexion and abduction (measured in standing), elbow flexion and extension (in supine), and forearm pronation-supination and wrist flexion-extension (in sitting). Movements will first be demonstrated on the unaffected limb, then performed with the affected limb. Active ROM values will be recorded. Each movement will be measured three times, and the mean value in degrees will be documented. Measurements will follow Kendall-McCreary criteria to ensure standardization and accuracy.
Muscle Strength Assessment | Baseline and after 8-weeks
  Muscle strength of shoulder flexion-abduction, elbow flexion-extension, forearm pronation-supination, and wrist flexion-extension will be assessed before and after treatment using a hand-held dynamometer (HOGGAN microFET2). A towel will be placed between the limb and device to ensure full contact and minimize sensitivity caused by surface hardness. The "make method," accepted for pediatric use, will be applied: the physiotherapist will ask the child to push maximally against the fixed device. The test will first be demonstrated on the unaffected limb. Two practice trials will be conducted on the affected side to ensure comprehension, followed by three test measurements. A rest interval will be given between trials. The mean of the three tests will be recorded in kilograms (kg).

SECONDARY OUTCOMES:
Quality of Upper Extremity Skills Test-QUEST | Baseline and after 8-weeks
  The Quality of Upper Extremity Skills Test (QUEST) is designed to assess upper extremity movement quality and hand function in children with cerebral palsy. It includes subtests for dissociated movements, grasp, weight-bearing, protective extension, hand function rating, spasticity grading, and cooperation. Each item is scored on a 3-point scale (0-2), based on whether the movement is successfully performed. The total score reflects the functional quality of the affected upper limb. The administration time is approximately 20-30 minutes.
ABILHAND- Kids | Baseline and after 8-weeks
  ABILHAND-Kids is a functional scale used to assess manual ability in children with cerebral palsy and other pediatric neurological disorders. It supports treatment planning and goal setting by evaluating the child's ability to perform daily activities requiring hand use. The scale consists of 21 items, most involving bimanual tasks, and measures the perceived difficulty of these activities as reported by parents. Each item is rated on a 3-point ordinal scale: 0 = impossible, 1 = difficult, and 2 = easy. The scale provides insight into hand performance in self-care tasks from the caregiver's perspective.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, ZEYTİNBURNU, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adiguzel H, Kirmaci ZIK, Gogremis M, Kirmaci YS, Dilber C, Berktas DT. The effect of proprioceptive neuromuscular facilitation on functional skills, muscle strength, and trunk control in children with cerebral palsy: A randomized controlled trial. Early Hum Dev. 2024 May;192:106010. doi: 10.1016/j.earlhumdev.2024.106010. Epub 2024 Apr 15. PMID 38653163
- [Background] Abd-Elmonem AM, Ali HA, Saad-Eldien SS, El-Nabie WAA. Efficacy of plyometric exercises on upper extremity function, selective motor control and hand grip strength in children with unilateral cerebral palsy: A randomized controlled study. Physiother Res Int. 2024 Jan;29(1):e2061. doi: 10.1002/pri.2061. Epub 2023 Nov 3. PMID 37922449